CLINICAL TRIAL: NCT02740322
Title: Validation of the Hum Test, a Simple and Reliable Alternative to the Weber Test
Brief Title: Validating the Hum Test
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution and no subjects enrolled
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-00102
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Hearing Loss
Keywords: Hum Test, Weber test, audiogram
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hum Test (Other): To examine and compare the Hum Test, Weber Test, and audiogram in their ability to detect and identify hearing loss, hearing loss will be simulated with the use of ear plugs (mimicking conductive hearing loss). Subjects will serve as their own control as these tests will be conducted with and without ear plugs.
  Interventions: Procedure: Hum Test; Procedure: Weber Test; Device: Audiogram

INTERVENTIONS:
Procedure: Hum Test — The subject will be brought into an exam room. The subject will then be asked to hum for a few seconds in a low pitch. They will then be asked if the nose was heard more so in one ear compared to the other. The subject will then be asked to hum for a few seconds in a high pitch. They will then be asked again if the noise was heard more so in one ear compared to the other.
Procedure: Weber Test — Using a 512 Hz tuning fork, the tuning fork will be vibrated and placed on the subject's glabella (forehead landmark). The subject will then be asked if the vibration was heard more so in one ear compared to the other.
Device: Audiogram — A standard audiogram will be administered by an audiologist.

SUMMARY:
The sensitivity and specificity of the Hum Test is being investigated in it's ability to detect conductive hearing loss. The hum test is simply elicited by asking the subject to hum to him or herself for a few seconds at both a high and low pitch that is comfortable for the subject. The subject is then asked if the hum was heard on one side more than the other (left or right), or if the sound was equal on both sides. To simulate conductive hearing loss, ear plugs will be placed in one of the subject's ears. We will elicit the hum test as well as the standard Weber test and audiogram across two conditions, with an ear plug and without an ear plug. From this, it is hoped to assess how the Hum Test compares to the audiogram (gold standard) in detecting conductive hearing loss as well as how it compares to the standard Weber test. If the Hum Test demonstrates strong sensitivity and specificity in detecting conductive hearing loss, it could have application as being utilized as an alternative to the standard Weber test, or in a setting where a formal physical examination may not yet be possible but where the etiology of a patient's hearing change could be quickly assessed remotely and thus the urgency of intervention/ consultation could then be determined.

DETAILED DESCRIPTION:
It is presumed that the Hum Test works similarly to the Weber Test, where bone conduction of the skull is elicited to determine if a change in hearing is conductive or sensorineural in nature. Because the hum test is frequently employed in clinical practice yet its validation has yet to be demonstrated, investigation is warranted.

To examine and compare the Hum Test, Weber Test, and audiogram in their ability to detect and identify hearing loss, hearing loss will be simulated with the use of ear plugs (mimicking conductive hearing loss). Subjects will serve as their own control as these tests will be conducted with and without ear plugs.

Study data will be maintained using an online, password protected storage system. No identifiable information will be collected or stored (i.e. name, DOB, etc.). Limited demographic information will be collected for analysis purposes such as age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Subjective normal hearing and no previous complaints or history of hearing problems or otologic disorders
* Subjects will be NYU medical students, NYU resident physicians, or patients from the Long Island Cochlear Implant Center

Exclusion Criteria:

* Has not had a URI (assessed by asking patient if they have had fever, cough, sore throat, nasal congestion, or runny nose) within one month of study session

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The correlation of the results between the Hum Test and the Audiogram | 30 minutes
  The Hum test will measure a subject's ability to hear a high pitch and a low pitch in each ear. The Audiogram will measure a subject's hearing threshold at various frequencies.
The correlation between the Hum Test and the Weber Test | 30 Minutes
  The Weber Test will measure a subject's ability to hear vibrations in both ears.

CONTACTS AND LOCATIONS:
Overall Officials: Erich Voigt, MD, Principal Investigator — NYU Langone Health